CLINICAL TRIAL: NCT07051174
Title: Minimally Invasive Micro Sclerostomy System - Long- Term Follow-Up Extension Study
Brief Title: The Minimally Invasive Micro Sclerostomy (MIMS®) System is Intended for the Reduction of Elevated Intraocular Pressure (IOP): The Minimally Invasive Micro Sclerostomy (MIMS®) System is Intended for the Reduction of Elevated Intraocular Pressure (IOP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMS EEU-3
Record Dates: First submitted 2025-05-28; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm: MIMS® Minimally Invasive Trabeculostomy in OAG Patients (36-Month Follow-Up) (Experimental): This follow-up extension study is aimed to monitor the long-term IOP-lowering performance/efficacy and safety of the MIMS® procedure in open angle glaucoma eyes.
  Interventions: Diagnostic Test: MIMS

INTERVENTIONS:
Diagnostic Test: MIMS — This study is an extension follow up study conducted in continuation of the prior MIMS® study (see: STUDY ID: MMS EEU-1), in which the long-term (i.e., 28, 36, 42 months) clinical outcomes of Minimally Invasive Micro Sclerostomy System [MIMS® System] [CE Marked device] are evaluated.

SUMMARY:
No new investigational device is used in this study. This study is an extension follow up study conducted in continuation of the prior MIMS® study (see: STUDY ID: MMS EEU-1), in which the long-term (i.e., 28, 36, 42 months) clinical outcomes of Minimally Invasive Micro Sclerostomy System [MIMS® System] [CE Marked device] are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years to ≤ 85 years old
* Subject who underwent either standalone MIMS® surgery or MIMS® surgery in combination with phacoemulsification, in continuation of the previous clinical investigation with the MIMS® device (see: STUDY ID: MMS EEU-1), and surgery was performed not earlier than 2 years from enrollment
* Subject who is considered complete success (i.e., 20% or greater reduction in IOP from Baseline on no medications) and qualified success (i.e., 20% or greater reduction in IOP from Baseline on the same or less number of medications) or failure with IOP >21mmHg with no medications at 1 year post MIMS® surgery (see: STUDY ID: MMS EEU-1)
* Subject who is able and willing to attend all scheduled assessments
* Subject understands and signs the informed consent

Exclusion Criteria:

* Subject who was considered failure at 1 year after the MIMS® surgery
* Any subject with major protocol deviation from the prior MIMS® study (ID: MMS EEU-1)
* Other secondary glaucoma (such as neovascular, uveitic, lens-induced, trauma-induced, or glaucoma associated with increased episcleral venous pressure) in the study eye, since the MIMS® surgery in the study eye
* Any ocular disease in the study eye such as severe dry eye, active proliferative retinopathy, ICE syndrome, epithelial or fibrous down growth, and ocular pathology that may interfere with accurate IOP measurements
* Any ocular surgery since the MIMS® surgery in the study eye
* Severe trauma in the study eye since the MIMS® surgery in the study eye
* Current participation or participation in another investigational drug or device clinical trial within the last 30 days before enrollment in the study
* Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Observed IOP at Long- Term ( >2 Years) post-MIMS® surgery: | 28 +/-3 months post-MIMS® surgery 36 +/-3 months post-MIMS® surgery 42 +/-3 months post-MIMS® surgery
  • IOP will be measured for subjects who have completed the MIMS® surgery and no earlier than 2 years from the procedure.

SECONDARY OUTCOMES:
• IOP Levels at the following time points: | 28 +/-3 months post-MIMS® surgery 36 +/-3 months post-MIMS® surgery 42 +/-3 months post-MIMS® surgery
  IOP will be measured for subjects who have completed the MIMS® surgery and assessed at least one of the following visits (the data from more than one visit will be also collected):
  28 +/-3 months post-MIMS® surgery 36 +/-3 months post-MIMS® surgery 42 +/-3 months post-MIMS® surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Malayan, Yerevan, Armenia